CLINICAL TRIAL: NCT07078552
Title: Research on Precision Diagnosis and Treatment Decision of Common Eye Diseases Based on Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1035
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Congenital Ptosis
Keywords: Congenital Ptosis; levator function
MeSH Terms: interventions — BPESC1 lncRNA, human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- congenital ptosis
  Interventions: Other: ptosis

INTERVENTIONS:
Other: ptosis — no intervention

SUMMARY:
The goal of this observational study is to investigate the clinical features of congenital ptosis in children by analyzing eyelid movement captured through smartphone videos. The main question it aims to answer is:

Can video-based eyelid measurements and levator muscle function grading provide useful guidance for the treatment of congenital ptosis in children?

Participants are children diagnosed with congenital ptosis. Their blinking behavior will be recorded using a smartphone, and eyelid morphology and muscle strength will be assessed from the video data.

DETAILED DESCRIPTION:
In this study, we developed a two-module system for the evaluation of congenital ptosis in children based on smartphone video recordings. The first module performs morphological measurements of eyelid parameters (e.g., palpebral fissure height, margin reflex distance) extracted from blink videos. The accuracy of this module was assessed through agreement analysis between automated measurements and manual measurements performed by clinicians.

The second module focuses on levator function grading. The automated grading results were compared against clinical assessments by senior oculoplastic specialists, which served as the gold standard, to evaluate the model's accuracy. Additionally, we compared the model's performance to that of junior ophthalmology residents to assess the system's clinical assistive value in real-world scenarios.

Based on these modules, we developed a smartphone-based application for remote ptosis assessment. A multi-center clinical validation study was designed to evaluate the feasibility, consistency, and generalizability of the system in different clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* participants aged ≤18 years with compliance during video recording. Congenital ptosis diagnosis mandated documented symptom onset within the first year of life and bilateral or unilateral MRD1 of < 2.5 mm

Exclusion Criteria:

* acquired ptosis, myasthenia gravis, Marcus Gunn syndrome, eyelid deformities, or prior ophthalmic surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inclusion criteria required participants aged ≤18 years with compliance during video recording. Congenital ptosis diagnosis mandated documented symptom onset within the first year of life and bilateral or unilateral MRD1 of < 2.5 mm. Healthy controls exhibited age-appropriate ocular development without eyelid abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
levator function testing | One-time assessment; results available within 1 week of data collection.

CONTACTS AND LOCATIONS:
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China